CLINICAL TRIAL: NCT01769924
Title: Effect of A Reduction in Glomerular Filtration Rate After Nephrectomy on Arterial Stiffness (EARNEST)
Brief Title: A Prospective UK Multicentre Study of Kidney Donors
Acronym: EARNEST
Status: Completed | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: British Heart Foundation (Other); University Hospital Birmingham NHS Foundation Trust (Other); North Bristol NHS Trust (Other); University Hospitals Coventry and Warwickshire NHS Trust (Other); St. George's Hospital, London (Other); Glasgow Western Infirmary (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Jonathan N. Townend, Consultant Cardiologist and Honorary Reader in Cardiology, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: A092761
Record Dates: First submitted 2013-01-08; First posted 2013-01-17 (Estimated); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Living Kidney Donors
Keywords: Kidney donors; Arterial stiffness; Blood pressure; Nephrectomy
MeSH Terms: interventions — Nephrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, serum and plasma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Live kidney donors: Nephrectomy
  Interventions: Other: Nephrectomy
- Healthy controls: Who also meet criteria to donate a kidney

INTERVENTIONS:
Other: Nephrectomy — Nephrectomy for the purposes of living kidney donation
  Groups: Live kidney donors

SUMMARY:
Studies of patients with established kidney disease, even when this is mild, appear to show that they are at high risk of heart failure, stroke and sudden cardiac death. This may be because kidney disease causes stiffening of the arteries in the body which means that the heart and brain are damaged by high blood pressure. By studying patients before and after the removal of a kidney (uni-nephrectomy) for transplantation the investigators will find out for the first time in man the effect of an isolated reduction in kidney function on the structure and function of the cardiovascular system.

DETAILED DESCRIPTION:
HYPOTHESIS

In living kidney donors, reduction in GFR post-nephrectomy results in:

1. A pressure-independent increase in aortic stiffness (aPWV)
2. An increase in peripheral and central blood pressure

EXPERIMENTAL DETAILS AND DESIGN OF PROPOSED INVESTIGATION We propose a prospective, longitudinal parallel group study of 200 kidney donors and 200 controls to be recruited over two years and followed up over one year.

Subjects: The only inclusion criterion is that subjects will be scheduled for nephrectomy for the purpose of kidney donation. Subjects will be recruited from centres, chosen because of their high numbers of live donor transplants and strength in vascular research.

Controls: We will recruit a carefully matched series of control patients from the same living donor clinics at which subjects are identified, who after screening are found to be fit for donation but do not proceed to surgery.

Exclusion criteria for both subjects and controls: These will be the current nationally set exclusion criteria for donors and will include diabetes mellitus, any history of cardiovascular or pulmonary disease, evidence of hypertensive end-organ damage, LV dysfunction (EF < 40%) and atrial fibrillation.49

Primary endpoint: Change in aPWV at 12 months adjusted for mean arterial pressure and heart rate at time of measurement compared with controls.

Secondary endpoints: Change in ambulatory blood pressure, AIx, central aortic pressure and urinary ACR compared with controls.

Secondary analysis: Change in endpoints will be analysed according to baseline GFR, change in GFR, pre-donation hypertension and ethnic group.

Investigations:

The following investigations will be performed in all subjects and controls at baseline (<6 weeks pre-donation) and 1 year post-donation. Subjects and controls will undergo routine follow up by the renal team with no alteration to normal care. No restrictions will be made to the introduction of any treatment including anti-hypertensive drugs. At baseline BMI, blood pressure and heart rate will be recorded. Routine haematological and biochemical parameters including lipids will be recorded. The following additional parameters will be determined:

1. Arterial stiffness: A Sphygmocor device will be used to measure parameters including aPWV, AIx and central aortic pressure.
2. Spot urine samples will be collected for measurement of ACR.
3. Clinic blood pressure
4. 24-hour ambulatory blood pressure studies (24h ABPM)
5. Isotope GFR for kidney donors will be measured using the renal clearance of 51Cr EDTA50, in keeping with national recommendations. Kidney function in controls will be estimated using MDRD eGFR to minimise radiation exposure and cost.

STATISTICS The original recruitment target was 800 patients. Power calculations used a SD of 1.0 m/s in aPWV and 10 mm Hg in blood pressure and a sample size of 800 patients (control and donors, 400 subjects each). This gives 80% power to detect a difference of 0.22 m/s or 2.2 mm Hg for aPWV and blood pressure allowing for 9% drop out. This is a 2-sided t test at the 2.5% significance level. During the study it was apparent the original recruitment target would not be met therefore a new sample size was calculated.

New power calculations:

Using a SD of 1.0m/s in aPWV and a sample size of 400 patients (control and donors, 200 subjects each). This gives a 92% power to detect a difference of 0.4m/s for aPWV and 4mm Hg for blood pressure allowing for 15% drop out (alpha at 5%). This is a 2-sided t test at the 2.5% significance level. Following this we aimed for a sample size of 400 patients (200 controls and 200 donors) for determination of the primary outcome of PWV in both groups.

ELIGIBILITY:
Inclusion Criteria:

* A donor group will be recruited from all patients undergoing donor nephrectomy.
* A contemporaneous control group will be recruited from clinics, advertisements within and outside the institutions and from any local volunteer databases.

Exclusion Criteria:

* These will be the same for donors and controls. The current nationally set exclusion criteria for donors include age/glomerular filtration rate (GFR) cutoff, diabetes mellitus, any history of cardiovascular or pulmonary disease, evidence of hypertensive end-organ damage, known left ventricular dysfunction (including ejection fraction < 40%) and atrial fibrillation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Aortic Pulse Wave Velocity (aPWV) adjusted for mean arterial pressure and heart rate | 12 months

SECONDARY OUTCOMES:
Clinic blood pressure | 12 months
Number of patients newly diagnosed with hypertension | 12 months
  As defined by commencement of antihypertensive therapy
Augmentation index (AIx) | 12 months
Central blood pressure | 12 months
  Central haemodynamics
N-terminal prohormone of brain natriuretic peptide (NT-proBNP) | 12 months
Urinary albumin: creatinine ratio (ACR) | 12 months
24 hr Ambulatory Systolic Blood Pressure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: John Cockcroft, PhD, Study Chair — Cardiff; Ian B Wilkinson, Study Director — Cambridge Heart Inc.; Jonathan N Townend, Principal Investigator — Birmingham
Locations (1):
- University Hospital Birmingham NHS Foundation Trust, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moody WE, Tomlinson LA, Ferro CJ, Steeds RP, Mark PB, Zehnder D, Tomson CR, Cockcroft JR, Wilkinson IB, Townend JN. Effect of A Reduction in glomerular filtration rate after NEphrectomy on arterial STiffness and central hemodynamics: rationale and design of the EARNEST study. Am Heart J. 2014 Feb;167(2):141-149.e2. doi: 10.1016/j.ahj.2013.10.024. Epub 2013 Nov 6. PMID 24439974
- [Derived] Price AM, Greenhall GHB, Moody WE, Steeds RP, Mark PB, Edwards NC, Hayer MK, Pickup LC, Radhakrishnan A, Law JP, Banerjee D, Campbell T, Tomson CRV, Cockcroft JR, Shrestha B, Wilkinson IB, Tomlinson LA, Ferro CJ, Townend JN; EARNEST investigators. Changes in Blood Pressure and Arterial Hemodynamics following Living Kidney Donation. Clin J Am Soc Nephrol. 2020 Sep 7;15(9):1330-1339. doi: 10.2215/CJN.15651219. Epub 2020 Aug 25. PMID 32843374